CLINICAL TRIAL: NCT04764097
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled Trial to Determine the Effect of Dapagliflozin 10mg Once Daily on Cardiovascular Outcomes in Haemodialysis for Patients With End Stage Renal Disease (ESRD)
Brief Title: Dapagliflozin Effect on Cardiovascular Outcomes in Haemodialysis for End Stage Renal Disease
Acronym: DECODED
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding and similar competing study being conducted in Europe.
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, David Foo Chee Guan, Adjunct Associate Professor, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TTSH-DECODED
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Cardiovascular Diseases; End Stage Renal Disease
Keywords: Cardiovascular Outcomes; Renal Disease; Dapagliflozin; SGLT2 Inhibitor
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Failure, Chronic; Kidney Diseases | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Randomised (1:1) to either Dapaglifozin 10mg or placebo.
Who Masked: Participant, Investigator
Masking Description: Double-blinded clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin, Oral Tablet,10mg, od, 24 months.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo, Oral Tablet, od, 24 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — SGTL2 Inhibitor
  Arms: Dapagliflozin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study aims to study SGLT2 inhibitors in patients who are undergoing haemodialysis for end stage renal disease and established ASCVD, to examine the safety and clinical outcomes, consisting of a composite of non-fatal stroke, non-fatal myocardial infarction, or cardiovascular death as the primary outcome. The key secondary composite outcome was all cause death or hospitalization for unstable angina.

DETAILED DESCRIPTION:
Cardiovascular disease accounts for more than 50% of end-stage renal disease (ESRD) deaths. The reported cardiovascular death rates in patients receiving dialysis are substantially higher than in the general population. Cardiovascular mortality in ESRD is particularly high after acute myocardial infarction, but it is also elevated in ESRD patients with other forms of atherosclerotic vascular disease (eg, chronic coronary artery disease, strokes, transient ischemic attacks, and peripheral arterial disease). Left ventricular hypertrophy and dilation are associated with increased cardiovascular mortality, as is congestive heart failure. One of the major reasons for such high cardiovascular mortality in ESRD is the large burden of cardiovascular disease present in patients with chronic artery disease before renal replacement therapy.

SGLT2 inhibitors have demonstrated benefits in reduction of major adverse cardiac events and heart failure hospitalisation in phase 3 randomised controlled trials. In addition, several recent clinical publications have also indicated renal benefits in patients with chronic renal impairment (eGFR >30ml/min).

The primary SGLT2 inhibition predominantly occurs at the proximal tubules of kidneys. The mechanistic benefits postulated (other than serum glucose lowering) included SGL2i mediated naturesis and glucosuria. Independent of this class's effects at the renal level, SGL2i possibly affect cardiac metabolism (in animal studies), with reverse adverse cardiac remodelling by switching myocardial substrate utilization from glucose toward oxidation of fatty acids, ketone bodies and branch-chained amino acids. Such improvement in cardiac metabolism may attenuate myocardial ischemia, improve cardiac haemodynamics and reduce overall cardiac mortality, either independent of or synergistic with SGLT2 inhibition at the kidney level.

Currently, there is a gap in knowledge and paucity of safety, efficacy and clinical outcomes data for the use of SGLT2 inhibitors in patients who are undergoing haemodialysis for end stage renal disease and established ASCVD.

This study aims to study SGLT2 inhibitors in this population and examine the safety and clinical outcomes, consisting of a composite of non-fatal stroke, non-fatal myocardial infarction, or cardiovascular death as the primary outcome. The key secondary composite outcome was all cause death or hospitalization for unstable angina.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Female or male aged ≥ 21 years.
* Undergoing haemodialysis for end stage renal disease regardless of cause and previous cardiac events.

Exclusion Criteria:

* Diagnosis of Type 1 diabetes mellitus.
* Pregnant or planning pregnancy or breast-feeding patients.
* Any clinical condition that would jeopardize patient safety while participating in this clinical trial.
* Intake of an investigational drug or participating in another clinical trial involving an investigational drug.
* Life limiting disease other than ESRD with life expectancy estimated to be less than 12 month.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Subjects included in the composite endpoint of cardiovascular death, myocardial infarction or ischemic stroke (time to first or recurrent event). | Up to 3 years
  Data will be derived from 3 monthly telephone follow-up and 6monthly physical site visits and events are documented in eCRF

SECONDARY OUTCOMES:
Subjects included in the composite endpoint of all-cause death or hospitalization for unstable angina (time to first or recurrent event). | Up to 3 years
  Data will be derived from 3 monthly telephone follow-up and 6monthly physical site visits and events are documented in eCRF

OTHER OUTCOMES:
Safety and tolerability will be assessed from overall adverse events, serious adverse events, adverse events of special interest | Up to 3 years
  The assessment will include an evaluation of the incidence of adjudicated hyperkalemia, diabetic ketoacidosis, thromboembolic event, genital infections, bone fractures,amputation, liver injury etc.Data will be derived from 3 monthly telephone follow-up and 6monthly physical site visits and events are documented in eCRF

IPD SHARING:
Plan to Share IPD: No